CLINICAL TRIAL: NCT04342260
Title: Improving Quality of Life After Thoracic Surgery Using Patient-Reported Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Thoracic Surgery Foundation (Unknown); American College of Surgeons (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: LCCC1945
Record Dates: First submitted 2020-03-24; First posted 2020-04-10 (Actual); Results first posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-01

CONDITIONS: Thoracic Surgery
Keywords: Patient-Reported Outcomes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Monitoring (Experimental): Clinicians will receive symptom alerts if the survey suggests increased or worsening symptoms.
  Interventions: Other: Active Monitoring
- Passive Monitoring (Active Comparator): Clinicians will not receive any symptom alerts.
  Interventions: Other: Passive Monitoring

INTERVENTIONS:
Other: Active Monitoring — The participants randomized to active symptom monitoring will have alerts sent to their clinicians when their PRO symptom scores exceed baseline postoperative scores (when discharge day scores are available) by 2 points or more, or when 'severe' or 'very severe' symptoms are reported.
  Arms: Active Monitoring
Other: Passive Monitoring — Participants randomized to the passive PRO monitoring arm will complete the same PROs as participants in the active monitoring arm, but will not have alerts sent to their clinician.
  Arms: Passive Monitoring

SUMMARY:
This study is designed to test if patient-reported outcomes with automated reporting to clinicians for remote monitoring of postoperative symptoms is feasible and improves quality of life, health outcomes, and service utilization in thoracic surgery patients. Patients undergoing thoracic surgery will be asked to self-report symptoms for remote monitoring by their care team.

DETAILED DESCRIPTION:
This is a single center, randomized feasibility study. A total of 140 patients undergoing thoracic surgery will be prospectively enrolled and randomized in a 1:1 ratio to one of two arms. All participants will complete patient-reported outcome (PRO) symptom monitoring. The two arms are 1) active symptom monitoring and 2) passive symptom monitoring. The participants randomized to active symptom monitoring will have alerts sent to their clinicians when their PRO symptom scores exceed baseline postoperative scores (when discharge day scores are available) by 2 points or more, or when 'severe' or 'very severe' symptoms are reported. Participants randomized to the passive PRO monitoring arm will complete the same PROs as participants in the active monitoring arm, but will not have alerts sent to their clinician. All participants will be administered survey instruments to assess quality of life, satisfaction, and health history. In addition, a subset of up to 40 participants will be chosen at 2 months postoperatively to complete a semi-structured interview about their postoperative symptom reporting experience.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* English speaking
* Able and willing to complete web-based symptom survey
* Be presenting for inpatient thoracic surgery

Exclusion Criteria:

* Not completing planned surgery within 3 months of obtaining informed consent
* Diagnosis of esophageal cancer
* Inability to read and speak English
* Presenting for a day surgery
* Presenting for foregut surgery (e.g. paraesophageal hernia repair)
* Dementia, altered mental status, or any psychiatric condition that would prohibit the understanding or rendering of informed consent.
* Current incarceration
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2020-04-30 (Actual); Primary Completion 2023-11-10 (Actual); Study Completion 2023-11-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gita Mody, MD, MPH, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
No plans as of now to make IPD available to other researchers.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients undergoing major thoracic surgery within the Multidisciplinary Thoracic Surgery Program at the University of North Carolina at Chapel Hill between April 2020 and June 2021 who met the inclusion criteria were invited to participate in this study.
Pre-assignment Details: Eligible patients who enrolled were assigned to study arms at the time of enrollment in a 1:1 ratio using block randomization with blocks of 20 participants (patients).
Period: Overall Study
Arm/Group | Active Monitoring | Passive Monitoring
Started | 56 | 57
Started ePROs | 50 | 49
Completed ePROs | 47 | 45
Completed | 28 | 30
Not Completed | 28 | 27

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Monitoring | Passive Monitoring | Total
Number analyzed (Participants) | 56 | 57 | 113
Age, Customized [Count of Participants; unit: Participants]
  <18 years | 0 | 0 | 0
  18-65 years | 38 | 27 | 65
  >65 years | 18 | 29 | 47
  Unknown | 0 | 1 | 1
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 32 | 38 | 70
  Male | 24 | 18 | 42
  Unknown | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 51 | 54 | 105
  Unknown or Not Reported | 3 | 3 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 39 | 43 | 82
  Black | 11 | 9 | 20
  Other | 6 | 4 | 10
  Unknown | 0 | 1 | 1
Region of Enrollment [Number; unit: number of participants]
  United States | 56 | 57 | 113

OUTCOME MEASURES:

1. Primary Outcome: Quality of Life at 12 Months
Description: Quality of Life (QOL) will be measured by the EORTC (European Organisation for Research and Treatment of Cancer) Quality of Life Questionnaire Core-30 (EORTC QLQ-C30) version 3.0 and reported as a score on a scale from 0 to 100 with a higher score being a better QOL.
Time Frame: 12 months post-discharge
Population: Intent to treat population.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Monitoring | Passive Monitoring
Number analyzed (Participants) | 50 | 49
units on a scale | 80.97 (17.06) | 84.02 (16.58)

2. Primary Outcome: Lung Cancer Specific Quality of Life at 12 Months
Description: Lung cancer specific Quality of Life will be measured by the EORTC (European Organisation for Research and Treatment of Cancer) Quality of Life Questionnaire Lung Cancer-13 (EORTC QLQ-LC13) supplement and reported as a score from 0 to 100 with a higher score being worse symptoms
Time Frame: 12 months post-discharge
Population: Intent to treat population.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Monitoring | Passive Monitoring
Number analyzed (Participants) | 50 | 49
units on a scale
  Pain in chest | 15.48 (27.94) | 9.52 (17.82)
  Pain in arm or shoulder | 21.43 (26) | 10.71 (22.32)
  Pain in other parts | 30.95 (32.62) | 21.43 (28.99)
  Peripheral neuropathy | 26.19 (34.38) | 13.1 (20.96)
  Dyspnea | 20.09 (22) | 23.81 (24.51)
  Coughing | 22.62 (24.09) | 30.95 (22.09)

3. Primary Outcome: PRO Symptom Monitoring Surveys Completed at 3 Months
Description: The percentage of subjects who completed symptom surveys out of delivered symptom surveys.
Time Frame: 3 months post-discharge
Population: Intent to treat population.
Measure: Number; unit: percentage of participants completed
Arm/Group | Active Monitoring | Passive Monitoring
Number analyzed (Participants) | 50 | 49
percentage of participants completed | 61.1 | 50.30

4. Primary Outcome: PRO Symptom Monitoring Alerts Resulting in a Clinician Response at 3 Months
Description: The percentage of survey alerts that generate a clinician response will be calculated.
Time Frame: 3 months post-discharge
Population: Intent to treat
Measure: Number; unit: percentage of participants received aler
Arm/Group | Active Monitoring
Number analyzed (Participants) | 50
percentage of participants received aler | 64

5. Primary Outcome: Barriers and Facilitators of PRO Monitoring After Thoracic Surgery
Description: Barriers and facilitators of PRO monitoring after thoracic surgery will be assessed using qualitative methods. A subset of patients and caregivers participated in semi-structured interviews. Thematic analysis was used to identify determinants.
Time Frame: assessed at 2 months through 2 years post-discharge
Population: The subset of patients who completed semi-structured interviews included those from both the active and passive monitoring arms and were combined for thematic analysis. No calculations across or between groups were performed for qualitative analyses. Numbers represented here are the number of themes derived from the interviews.
Measure: Number; unit: Themes
Groups:
- Interview Subset: Subset of participant who completed semi-structured interviews.
Arm/Group | Interview Subset
Number analyzed (Participants) | 16
Themes
  Symptoms and physical functioning during surgical recovery were barriers to ePRO completion. | 1
  Access to required technology was a barrier to completing web-based ePROs for a few participants. | 1
  Participants reported ease of completing the ePRO assessments. | 1
  Patients preferred engagement on ePRO participation with the surgical care team. | 1
  Participants reported irrelevant or repeated ePRO monitoring questions. | 1
  Participants reported a lack of clarity on ePRO assessment integration with routine clinical care. | 1
  Participants reported increased awareness of their symptoms and recovery with ePRO use. | 1

6. Secondary Outcome: Readmission at 3 Months
Description: Readmission rates after thoracic surgery.
Time Frame: 3 months post-discharge
Population: Intent to treat
Measure: Count of Participants; unit: Participants
Arm/Group | Active Monitoring | Passive Monitoring
Number analyzed (Participants) | 50 | 49
Participants | 6 | 7

7. Secondary Outcome: Overall Survival at 12 Months
Description: Survival will be compared between arms using Cox proportional hazards regression model.
Time Frame: 12 months post-discharge
Population: Intent to treat
Measure: Count of Participants; unit: Participants
Arm/Group | Active Monitoring | Passive Monitoring
Number analyzed (Participants) | 50 | 49
Participants | 47 | 47

ADVERSE EVENTS:
Time Frame: This study protocol does not require Adverse Event reporting, only all-cause mortality up to12 months were reported.
Description: This study protocol does not require Adverse Event reporting, only unanticipated problems involving risks to study subjects or others (UPIRSO) refer to any incident, experience report is required.
Arm/Group | Active Monitoring | Passive Monitoring
All-Cause Mortality (participants affected / at risk) | 3/50 | 2/49
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-05): https://cdn.clinicaltrials.gov/large-docs/60/NCT04342260/Prot_SAP_000.pdf